CLINICAL TRIAL: NCT00003251
Title: A Pilot Study of Amifostine and Concomitant Cisplatin, Paclitaxel and Radiotherapy in Previously Irradiated, Recurrent Head and Neck Cancer
Brief Title: Amifostine Plus Chemotherapy and Radiation Therapy in Treating Patients With Advanced, Unresectable Head and Neck Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Illinois at Chicago (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Supportive Care
Other Study IDs: CDR0000066133; UIC-H-97-783; ALZA-UIC-H-97-783; NCI-V98-1389
Record Dates: First submitted 1999-11-01; First posted 2004-08-13 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2000-06

CONDITIONS: Drug/Agent Toxicity by Tissue/Organ; Head and Neck Cancer; Radiation Toxicity
Keywords: stage III nasopharyngeal cancer; stage IV nasopharyngeal cancer; recurrent nasopharyngeal cancer; stage III salivary gland cancer; stage IV salivary gland cancer; recurrent salivary gland cancer; salivary gland squamous cell carcinoma; high-grade salivary gland mucoepidermoid carcinoma; stage III lip and oral cavity cancer; stage IV lip and oral cavity cancer; recurrent lip and oral cavity cancer; stage III hypopharyngeal cancer; stage IV hypopharyngeal cancer; recurrent hypopharyngeal cancer; stage III laryngeal cancer; stage IV laryngeal cancer; recurrent laryngeal cancer; stage III paranasal sinus and nasal cavity cancer; stage IV paranasal sinus and nasal cavity cancer; recurrent paranasal sinus and nasal cavity cancer; stage III oropharyngeal cancer; stage IV oropharyngeal cancer; recurrent oropharyngeal cancer; stage III squamous cell carcinoma of the lip and oral cavity; stage III mucoepidermoid carcinoma of the oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV mucoepidermoid carcinoma of the oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; drug/agent toxicity by tissue/organ; radiation toxicity
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Head and Neck Neoplasms; Radiation Injuries; Nasopharyngeal Neoplasms; Salivary Gland Neoplasms; Mouth Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Oropharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Amifostine; Cisplatin; Paclitaxel; Radiotherapy

INTERVENTIONS:
Drug: amifostine trihydrate
Drug: cisplatin
Drug: paclitaxel
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses x-rays to damage tumor cells. Drugs, such as amifostine, may protect normal cells from the side effects of chemotherapy and radiation therapy.

PURPOSE: Phase I/II trial to study the effectiveness of amifostine plus cisplatin, paclitaxel, and radiation therapy in treating patients who have advanced unresectable head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the efficacy and role of amifostine as a cytoprotection agent with concurrent chemoradiotherapy in advanced, previously irradiated or metastatic head and neck cancer. II. Determine the toxicity and response to cisplatin, paclitaxel and radiation therapy in these patients. III. Determine the toxicity of amifostine in these patients.

OUTLINE: This is an open label study. Patients receive paclitaxel by continuous infusion on days 0-3. Amifostine IV is administered over 5 minutes on days 1-5. Radiation therapy is administered once daily on days 1-5. Cisplatin IV is administered on day 5. Patients receive no treatment on days 6-13. Treatment is repeated every 2 weeks for up to 7 courses in the absence of disease progression and unacceptable toxicity. Patients are followed monthly during the first year, every 2 months during the second year, then every 3 months thereafter.

PROJECTED ACCRUAL: This study will accrue 16-46 patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically documented metastatic or previously irradiated recurrent locoregional squamous cell or mucoepidermoid carcinoma of the head and neck Unresectable disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 OR Karnofsky 70-100% Life expectancy: Greater than 4 months Hematopoietic: WBC at least 3000/mm3 Platelet count at least 100,000/mm3 Granulocyte count at least 1500/mm3 Hepatic: Bilirubin no greater than 2.5 times normal SGOT and SGPT no greater than 2.5 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL Creatinine clearance at least 60 mL/min Other: No other significant infection No other medical or psychiatric illness Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 1 month since prior chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 3 months since prior radiotherapy (patients with recurrent disease) to head and neck region Surgery: Not speciified Other: At least 24 hours since antihypertensive medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 1997-12

CONTACTS AND LOCATIONS:
Overall Officials: Fred R. Rosen, MD, Study Chair — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago Health Sciences Center, Chicago, Illinois, United States